CLINICAL TRIAL: NCT05336383
Title: Phase II Study of Salvage Radiation Treatment After B-cell Maturation Antigen Chimeric Antigen Receptor T-cell Therapy for Relapsed Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1139; NCI-2022-03304 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm; Malignant Plasma Cell Neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation Therapy (Experimental): Radiation treatment will be to bony or soft tissue plasmacytomas in up to five radiation treatment fields to 10-20Gy (or equivalent dose in 2Gy fractions of 10-21Gy
  Interventions: Drug: Radiation Therapy

INTERVENTIONS:
Drug: Radiation Therapy — Given by Infusion

SUMMARY:
This study is a Phase II study to determine the preliminary safety and efficacy of salvage radiation treatment after BCMA CAR-T therapy in subjects with RRMM.

The study population will consist of subjects with RRMM previously treated with SOC BCMA CAR-T cell therapy with active disease on the D30+ PET or other imaging scan after CAR-T infusion. Patients who are planned for salvage chemotherapy less than 14 days after completion of radiation treatment will be excluded.

Radiation treatment will be to bony or soft tissue plasmacytomas in up to five radiation treatment fields to 10-20Gy (or equivalent dose in 2Gy fractions of 10-21Gy). Final dose, target, and technique are per treating radiation physician discretion within these guidelines.

Thirty patients will be enrolled. The co-primary endpoints are objective response rate (ORR) at 6 months and duration of response (DOR) among responders.

DETAILED DESCRIPTION:
Objectives

Primary Objective:

• The primary objective of the study is to evaluate the preliminary efficacy of salvage radiation therapy after BCMA CAR-T cell therapy in subjects with RRMM.

Secondary Objectives:

• Evaluate the safety of and other efficacy parameters of radiation treatment after BCMA CAR-T cell therapy in subjects with RRMM

Exploratory Objectives:

* Evaluate the immunophenotype and/or expression profile, and perform functional bulk and single cell analysis of CAR T cells, endogenous T cells as well as other immune cells in the blood, bone marrow and/or tumor tissue with BCMA CAR-T therapy and RT
* Evaluate changes in the levels of cytokines, chemokines, and soluble factors in the blood with BCMA CAR-T therapy and RT
* Evaluate changes in T cell receptor repertoire with BCMA CAR-T therapy and RT
* Evaluate gut microbiome of patients treated with BCMA CAR-T therapy and RT

ELIGIBILITY:
Inclusion criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF)
2. Subject is diagnosed with multiple myeloma
3. Subject previously received treatment with standard of care BCMA CAR-T cell therapy
4. Day 30 or later PET scan or other imaging scan after CAR-T infusion shows active disease
5. Subject has at least one myeloma lesion (plasmacytoma either in bone or soft tissue) that can be treated with radiation
6. Able to provide informed consent

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subjects in whom salvage chemotherapy is planned less than 14 days after the completion of radiation treatment
2. Subject is undergoing active treatment for another malignancy other than multiple myeloma
3. Pregnant women will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | through study completion, an average of 1 year
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma (Kumar, 2016)
Duration of response (DoR) among responders | through study completion, an average of 1 year
  Time from first documentation of response (PR or greater) to first documentation of progressive disease (PD) or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Penny Fang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org